CLINICAL TRIAL: NCT00248326
Title: The Genetic Basis of Atrial Fibrillation
Brief Title: The Genetic Basis of Atrial Fibrillation (AF)
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: EP Research funds (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0405107
Record Dates: First submitted 2005-11-02; First posted 2005-11-03 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; genetics; genetic polymorphisms
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients of the Cardiovascular Institute with known cardiac conditions and no history of atrial fibrillation.
- 2: Patients of the Cardiovascular Institute with known cardiac conditions and a history of atrial fibrillation.

SUMMARY:
The investigators' goal with this research is to:

1. Establish a clinical database and a DNA bank for 1000 individuals with AF and 1000 individuals without AF.
2. Directly test the hypothesis that known functional polymorphisms in the coding sequences and the promoter regions of cardiac genes (ion channels and genes known to affect survival in the setting of left ventricular dysfunction) predispose individuals to AF.

Over the past decade, advancing techniques and technologies for gene characterization have yielded significant clues as to the molecular mechanism of certain human heart rhythm disorders. The role of ion channel polymorphisms in subjects with AF is unknown. Similarly, it is also not known whether polymorphisms in other genes have an impact on the risk of AF.

The ability to characterize genomic "at-risk" profiles would have many potential benefits for patient care. Paramount among these is:

1. Increased oversight or intervention of at-risk subjects, which might prevent unnecessary morbidity and mortality due to AF.
2. Further insight into the pathogenesis of AF, which may lead to preventative or curative therapies.

DETAILED DESCRIPTION:
Atrial fibrillation (AF), a heart rhythm disorder, is a major health problem. As many as 3 million US persons are afflicted; this number is expected to rise significantly in coming decades because AF incidence is directly correlated with age. AF is significantly associated with cardiovascular morbidity and mortality.

Our goal with this research is to:

1. Establish a clinical database and a DNA bank for 1000 individuals with AF and 1000 individuals without AF.
2. Directly test the hypothesis that known functional polymorphisms in the coding sequences and the promoter regions of cardiac genes (ion channels and genes known to affect survival in the setting of left ventricular dysfunction) predispose individuals to AF.

Over the past decade, advancing techniques and technologies for gene characterization have yielded significant clues as to the molecular mechanism of certain human heart rhythm disorders. The role of ion channel polymorphisms in subjects with AF is unknown. Similarly, it is also not known whether polymorphisms in other genes have an impact on the risk of AF.

The ability to characterize genomic "at-risk" profiles would have many potential benefits for patient care. Paramount among these is:

1. Increased oversight or intervention of at-risk subjects, which might prevent unnecessary morbidity and mortality due to AF.
2. Further insight into the pathogenesis of AF, which may lead to preventative or curative therapies.

Subjects will be recruited from the patient pool of the Cardiovascular Institute (including the Comprehensive Heart Center and the PUH Outpatient Cardiology Clinic). For each subject enrolled, we will record demographic information; etiology and details of heart disease; family history of heart disease; non-cardiac medical history; physical exam findings; medicinal therapy; and results of prior cardiac testing (such as echocardiograms [Echo], gated blood pool scans of heart function [MUGAs], exercise stress tests [ESTs] cardiac catheterizations, and clinical electrophysiology studies [EP Studies]. Records will be maintained with identifiers in a locked file cabinet in the office of the Principal Investigator.

A blood sample of ~10 ml will be drawn from each participating subject on the day of enrollment. Blood samples will be drawn only once from each subject. There is no further follow up required for the subject. Blood will be sent to the University of Pittsburgh School of Medicine Cardiovascular Research Center where nucleated cells will be isolated from whole blood by centrifugation. DNA will be isolated from nucleated cells and stored at the Cardiovascular Research Center (on the 17th floor of the Biomedical Science Tower). All DNA samples will be coded to ensure confidentiality, and maintained in a locked freezer for the duration of the study (5 years). Samples will be destroyed if requested by the subject. Samples (blood and DNA) will be under the control of the Principal Investigator. The DNA samples will be used to identify polymorphisms in ion channel genes, as well as other genes that may be associated with an increased risk of AF. Genotyping of polymorphisms will be performed on the genomic DNA. The genomic DNA will be amplified by polymerase chain reaction method using gene-specific primers. For each polymorphism, genotype will be identified. We will determine the frequency of that genotype in our study population, and attempt to define significant associations with AF.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Able to give informed consent

Exclusion Criteria:

* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects must be patients of the UPMC Cardiovascular Institute who are under the medical care of UPMC cardiologists.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2005-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S. Schwartzman, MD, Principal Investigator — University of Pittsburgh/UPMC
Locations (1):
- University of Pittsburgh Medical Center/Comprehensive Heart Ctr., Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Gensini F, Padeletti L, Fatini C, Sticchi E, Gensini GF, Michelucci A. Angiotensin-converting enzyme and endothelial nitric oxide synthase polymorphisms in patients with atrial fibrillation. Pacing Clin Electrophysiol. 2003 Jan;26(1P2):295-8. doi: 10.1046/j.1460-9592.2003.00036.x. PMID 12687832
- [Background] Lai LP, Lin JL, Lin CS, Yeh HM, Tsay YG, Lee CF, Lee HH, Chang ZF, Hwang JJ, Su MJ, Tseng YZ, Huang SK. Functional genomic study on atrial fibrillation using cDNA microarray and two-dimensional protein electrophoresis techniques and identification of the myosin regulatory light chain isoform reprogramming in atrial fibrillation. J Cardiovasc Electrophysiol. 2004 Feb;15(2):214-23. doi: 10.1046/j.1540-8167.2004.03423.x. PMID 15028053
- [Background] Gaudino M, Andreotti F, Zamparelli R, Di Castelnuovo A, Nasso G, Burzotta F, Iacoviello L, Donati MB, Schiavello R, Maseri A, Possati G. The -174G/C interleukin-6 polymorphism influences postoperative interleukin-6 levels and postoperative atrial fibrillation. Is atrial fibrillation an inflammatory complication? Circulation. 2003 Sep 9;108 Suppl 1:II195-9. doi: 10.1161/01.cir.0000087441.48566.0d. PMID 12970232